CLINICAL TRIAL: NCT02528552
Title: A Multi-center, Randomized, Controlled, Double-blind Study That Evaluates a Low Level Laser Therapy Over-the-counter at Home Device, Theradome™ LH80 PRO vs a Sham Device, for Promoting Hair Growth in Males Diagnosed With Androgenetic Alopecia
Brief Title: Treatment of Androgenetic Alopecia in Males With Theradome™ LH80 PRO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradome, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR-PRC-001
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LH80 PRO (Active Comparator): Low level laser therapy
  Interventions: Device: LH80 PRO
- Sham device (Sham Comparator): No low level laser therapy
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: LH80 PRO
  Arms: LH80 PRO
Device: Sham Device
  Arms: Sham device

SUMMARY:
This is a prospective, randomized double-blind, multi-center study to evaluate the efficacy of low level laser therapy over-the-counter at home device Theradome LH80 PRO, compared to SHAM for promoting hair growth in males diagnosed with androgenetic alopecia, and a usability study to assess subject ability to self-assess hair loss and understanding use of the device.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be diagnosed with androgenetic alopecia with Norwood Hamilton hair loss scale of IIa, III vertex, IV and V.
* Subject must have Fitzpatrick skin type scale I to IV.
* Subject must be able to visit clinic site for baseline, 13 week and 26 week study visits and attend 2 visits by phone ( 6 and 19).
* Hair must be at least 1 inch in length. The hairstyle and length shall be the same for each site visit. Subjects are instructed to have their hair cut/styled 1-5 days in advance of a site visit.
* Be willing to undergo all study procedures including consent for global photographs of hair loss/growth and a 1 mm tattoo to mark the macrophotography site along the indicated transition area of the scalp between the hairline and the balding area of the vertex.
* Be willing to avoid use of wigs, hairpieces, and/or hair extensions during the study period.
* Ability to communicate effectively with study personnel.
* Agrees to abstain from use of any hair growth affecting oral or topical medication including over the counter and herbal medications, minoxidil, finasteride or dutasteride during the course of this study

Exclusion Criteria:

* History of taking Propecia or any other hair growth supplements for 12 months prior to enrollment.
* History of using Rogaine for 6 months prior to enrollment.
* Subject must have no previous hair transplant, cell treatment, micro needling, or any other treatment in the last 6 months in the scalp.
* Subject is currently suffering from an active autoimmune disease such as serum lupus erythematosus, or alopecia areata.
* Currently suffering from dermatologic condition in the treatment area or has a significant scar in the hair treatment area that, in the opinion of the investigator, will make hair growth difficult (such as systemic burns, etc).
* Subject has a sensitivity or allergy to tattoo ink.
* Clinically significant medical or psychiatric illness currently or within 30 days of study screening as determined by the investigator.
* Employed by sponsor, clinic site, or entity associated with the conduct of the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Hair growth | 26 weeks
  Determination of hair growth vs baseline through global photographic review by a blinded reviewer(s).
Quantitative Hair Growth | 26 weeks
  Change from baseline in non-vellus Terminal Hair count (≥ 30 μm) as measured with macrophotography (aka trichogram).

SECONDARY OUTCOMES:
Subject Self Assessment | 26 weeks
  Determination of subject ability to self-assess hair loss and correctly use the device via direct observation and use of diary.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Axis Clinical Tirals, Los Angeles, California
  - MedaPhase, Inc., Newnan, Georgia
  - NW Dermatology & Research Center, LLC, Portland, Oregon
  - Tennessee Clinical Research Center, Nashville, Tennessee